CLINICAL TRIAL: NCT02561533
Title: Immunohistochemical Detection of the BRAFV600E Mutation on Cytological Specimen in PTC
Brief Title: Detection of BRAF Mutation on FNAB From Papillary Thyroid Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristine Zøylner Rubeck, MD PhD-student, University of Aarhus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TIHCDBMTC1
Record Dates: First submitted 2015-09-17; First posted 2015-09-28 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Papillary Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BRAF immunohistochemistry (IHC) (Experimental)
  Interventions: Other: BRAF detection on fine needle aspiration biopsy (FNAB)

INTERVENTIONS:
Other: BRAF detection on fine needle aspiration biopsy (FNAB)

SUMMARY:
Immunohistochemical detection of the BRAF-V600E mutation on pre-operative fine needle aspiration biopsy (FNAB) from patients suspected for papillary thyroid carcinoma, using the mutation specific antibody VE1.

DETAILED DESCRIPTION:
The BRAF mutation is reported to be present in approximately 50% of papillary thyroid carcinomas (PTC). The mutation has been associated with poor prognosis and more advanced disease stage. Therefore, pre-operative detection of the BRAF-V600E mutation may be of clinical interest in order to individualize treatment of patients with BRAF positive PTC.

FNABs are performed immediately before the thyroid operation, and BRAF-V600E detection using VE1 is performed on clots. The VE1 stain is compared to the mutation status of the removed cancer or control tissue using the Cobas test.

ELIGIBILITY:
Inclusion Criteria:

* Bethesda system of reporting thyroid cytology (BSRTC) group 5-6 on pre-operative FNAB from the nodule (>1cm)
* Undergoing thyroid surgery (histology of index nodule)

Exclusion Criteria:

* Not undergoing thyroid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Immunohistochemical detection of BRAF mutation on fine needle aspiration biopsy (FNAB) | 1 day
  Mutations status correlated to histological diagnoses and mutation status on histological samples

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark